CLINICAL TRIAL: NCT03301090
Title: A Phase I Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of Co-administered MERS-CoV Antibodies REGN3048 and REGN3051 vs. Placebo in Healthy Adults
Brief Title: A Safety, Tolerability, Pharmacokinetics and Immunogenicity Trial of Co-administered MERS-CoV Antibodies REGN3048 and REGN3051
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-0109; HHSN272201500005I
Record Dates: First submitted 2017-09-14; First posted 2017-10-04 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2017-09-22

CONDITIONS: Corona Virus Infection
Keywords: Adults; Evaluate; Healthy; Immunogenicity; MERS-CoV; Pharmacokinetics; Phase I; Placebo; REGN MERS; Safety; Tolerability
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort A (Experimental): REGN3048+REGN3051 3 mg/kg (1.5 mg/kg of each mAb) single infusion IV, n=6; placebo IV, n=2
  Interventions: Other: Placebo; Biological: REGN3048; Biological: REGN3051
- Cohort B (Experimental): REGN3048+REGN3051 10 mg/kg (5 mg/kg of each mAb) single infusion IV, n=6; placebo IV, n=2
  Interventions: Other: Placebo; Biological: REGN3048; Biological: REGN3051
- Cohort C (Experimental): REGN3048+REGN3051 30 mg/kg (15 mg/kg of each mAb) single infusion IV, n=6; placebo IV, n=2
  Interventions: Other: Placebo; Biological: REGN3048; Biological: REGN3051
- Cohort D (Experimental): REGN3048+REGN3051 50 mg/kg (25 mg/kg of each mAb) single infusion IV, n=6; placebo IV, n=2
  Interventions: Other: Placebo; Biological: REGN3048; Biological: REGN3051
- Cohort E (Experimental): REGN3048+REGN3051 100 mg/kg (50 mg/kg of each mAb) single infusion IV, n=6; placebo IV, n=2
  Interventions: Other: Placebo; Biological: REGN3048; Biological: REGN3051
- Cohort F (Experimental): REGN3048+REGN3051 150 mg/kg (75 mg/kg of each mAb) single infusion IV, n=6; placebo IV, n=2
  Interventions: Other: Placebo; Biological: REGN3048; Biological: REGN3051

INTERVENTIONS:
Other: Placebo — Placebo
Biological: REGN3048 — REGN3048 is a fully monoclonal antibody (mAbs) which binds to the S protein of MERS-CoV.
Biological: REGN3051 — REGN3051 is a fully human monoclonal antibody (mAb) which binds to the S protein of MERS-CoV. It can reduce virus titers and ameliorate MERS-CoV-induced lung pathology when given post infection.

SUMMARY:
This is a Phase 1, first-in-human (FIH), single site, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics (PK), and immunogenicity of single ascending doses of a co-administered (1:1, w/w) combination of REGN3048 and REGN3051 mAb's, administered IV in healthy adult volunteers. Study duration of approximately 16 months. Approximately 48 evaluable subjects will be enrolled in the study, eight (8) subjects in each one of 6 sequential ascending IV dose cohorts. In each cohort, subjects will be randomized to receive mAb's REGN3048 and REGN3051 (6 subjects) or placebo (2 subjects). Primary Objective: To assess the safety and tolerability of REGN3048 and REGN3051 following co-administration of single, ascending IV doses of 1.5, 5, 15, 25, 50, and 75 mg/kg of each of the two mAb's.

DETAILED DESCRIPTION:
This is a Phase 1, first-in-human (FIH), single site, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics (PK), and immunogenicity of single ascending doses of a co-administered (1:1, w/w) combination of REGN3048 and REGN3051 mAb's, administered IV in healthy adult volunteers. Study duration of approximately 16 months. Approximately 48 evaluable subjects will be enrolled in the study, eight (8) subjects in each one of 6 sequential ascending IV dose cohorts. In each cohort, subjects will be randomized to receive mAb's REGN3048 and REGN3051 (6 subjects) or placebo (2 subjects). Primary Objective: To assess the safety and tolerability of REGN3048 and REGN3051 following co-administration of single, ascending IV doses of 1.5, 5, 15, 25, 50, and 75 mg/kg of each of the two mAb's. Secondary Objectives: 1) To assess the pharmacokinetic (PK) profiles of REGN3048 and REGN3051 following co-administration of single IV doses (1.5, 5, 15, 25, 50, and 75 mg/kg of each of the two mAb's); 2) To assess the immunogenicity of REGN3048 and REGN3051 following co-administration of single IV doses (1.5, 5, 15, 25, 50, and 75 mg/kg of each of the two mAb's)

ELIGIBILITY:
Inclusion Criteria:

All must be answered yes for the subject to be eligible for study participation

1. Informed consent understood and signed prior to initiation of any study procedures
2. Healthy male or healthy, non-pregnant, non-lactating female, meeting eligibility criteria as assessed by the clinicians listed on the FDA Form 1572
3. Willingness to comply and be available for all protocol procedures including inpatient confinement for about 3 days
4. Age between 18 and 45 years, inclusive on the day of infusion
5. Body Mass Index (BMI) of > or =18.5 and >or =30 kg/m2 and Weight > or = 50 kg (110 lbs) and < or = 100 kg (220 lbs)
6. In female subject of childbearing potential, a negative serum pregnancy test at screening and negative serum test within 24 hours prior to infusion Note: A woman is considered of childbearing potential unless post-menopausal (> or = 1 year without menses without other known or suspected cause and appropriately elevated FSH) or surgically sterilized via bilateral oophorectomy or hysterectomy
7. Females of childbearing potential and males agree to use acceptable contraception for the duration of the study Note: A highly effective method of birth control is defined as one that results in a low failure rate (i.e., less than 1 percent per year) according to the CDC criteria.30. These include progestin implants, intrauterine devices (IUDs), surgical (hysterectomy or tubal ligation; vasectomy) or abstinence. Use of methods with higher failure rate (such as progestin injectables, combined oral hormonal contraceptives, condoms, and diaphragms) will not be acceptable when used alone, but they could be considered, if used in combination with another method (for example, a female using combined oral contraceptives if her male partner is sterile, or if she and her non-sterile male partner use a double-barrier method), after consultation with the DMID MM. All males will be required to use a barrier method (condoms) for the duration of the study
8. Screening laboratory tests, are in the normal reference range with acceptable exceptions

   Notes:
   1. If urinalysis by dipstick is abnormal, a complete urinalysis with microscopic evaluation will be performed and the results will supersede the results of the dipstick for blood, glucose and protein.
   2. Menstruating females failing inclusion criteria due to a positive blood on urine test (dipstick or microscopic urinalysis) may be retested following cessation of menses. Do not exclude subjects with <5 RBC/HPF.
   3. Other laboratory values that are outside the range of eligibility but are thought to be due to an acute condition or due to collection or laboratory error may be repeated once.
9. Vital signs are within the acceptable range
10. Has adequate venous access for the infusion and blood collection
11. The urine drug screen is negative
12. Willing to abstain from alcohol consumption for a period of 2 days prior to and during the study
13. Available for follow-up for the duration of the study

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria are not eligible for participation.

All must be answered no for the subject to be eligible for study participation

1. History of a chronic medical condition that would either interfere with the accurate assessment of the objectives of the study or increase the risk profile of the subject.

   Note: Chronic medical conditions include diabetes; Asthma requiring use of medication in the year before screening; Autoimmune disorder such as lupus, Wegener's, rheumatoid arthritis, thyroid disease; Coronary artery disease; Chronic hypertension; History of malignancy except low-grade (squamous and basal cell) skin cancer thought to be cured; chronic renal, hepatic, pulmonary, or endocrine disease; myopathy, and neuropathy
2. History of severe allergic reaction of any type to medications, bee stings, food, or environmental factors or hypersensitivity or reaction to immunoglobulins.

   Note: Severe allergic reaction is defined as any of the following: anaphylaxis, urticaria, or angioedema
3. A marked baseline prolongation of QT/QTcF interval (e.g., repeated demonstration of a QTcF interval >450 milliseconds)
4. Clinically significant abnormal electrocardiogram at screening Note: Clinically significant abnormal ECG results include: complete left or right bundle branch block; other ventricular conduction block; 2nd degree or 3rd degree atrioventricular (AV) block; sustained ventricular arrhythmia; sustained atrial arrhythmia; two Premature Ventricular Contractions in a row; pattern of ST elevation felt consistent with cardiac ischemia; or any condition deemed clinically significant by a study investigator
5. Positive serology results for HIV, HBsAg, or HCV antibodies
6. Febrile illness with temperature >37.6°C 7 days prior to dosing
7. Pregnant or breastfeeding
8. Donated whole blood or blood products within 56 days prior to dosing or plans to donate blood prior to the last scheduled visit in the study (Day 121) Note: Blood products are defined as red blood cells, white blood cells, platelets or plasma)
9. Known allergic reactions to doxycycline or to any of the study product components present in the formulation or in the processing, as listed in the Investigator Brochure
10. Treatment with another investigational product within 30 days of dosing, including a drug, vaccine, biologic, device or blood product
11. Treatment with a monoclonal antibody at any time in the past or planned use during the study period
12. Receipt of antibody* or blood transfusion within 6 months of dosing or within 5 half-lives of the specific product given

    * Note: Tetanus Immune Globulin [TIG], Varicella-Zoster Immune Globulin [VZIG], Intravenous Immunoglobulin [IVIG], Intramuscular [IM] gamma globulin
13. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
14. Use of H1 antihistamines or beta-blockers within 5 days of dosing
15. Use of any prohibited medication within 30 days prior to study dosing or planned use during the study period Note: Prohibited medications include immunosuppressives (except nonsteroidal antiinflammatory drugs [NSAIDS]); immune modulators; oral corticosteroids (topical/intranasal steroids are acceptable); anti-neoplastic agents; any licensed biologic including monoclonal antibody or vaccine with the exception of licensed influenza vaccine during the flu season, which is allowed 7 days prior to dosing or 7 days after dosing
16. Any specific condition that in the judgment of the investigator precludes participation because it could affect subject safety
17. Plans to enroll or is already enrolled in another clinical trial that could interfere with safety assessment of the investigational product at any time during the study period Note: Includes trials that have a study intervention such as a drug, biologic, or device
18. Is a study site employee or staff who are paid entirely or partially by the NIAID Office of Clinical Research Resources (OCRR) contract for the DMID-funded trial Note: Site employees or staff include the PIs and sub-investigators or staff who are supervised by the PI or Sub-Investigators

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-01-19 (Actual); Study Completion 2019-01-19 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in abbreviated physical examination | Days 1-2
Changes from baseline in clinical safety laboratory values | From Day 2 up to Day 121
Changes from baseline in Electrocardiogram (ECG) parameters | 15 mins after infusion
Changes from baseline in Electrocardiogram (ECG) parameters | 24 hrs after infusion
Changes from baseline in symptom-directed physical examination | From Day 1 up to Day 121
Changes from baseline in vital signs | From Day 1 up to Day 121
The incidence of Adverse Events | From Day 1 up to Day 121
The incidence of treatment-emergent Serious Adverse Events | From Day 1 up to Day 121
The severity of Adverse Events assessed by toxicity grading criteria | From Day 1 up to Day 121
The severity of treatment-emergent Serious Adverse Events assessed by toxicity grading criteria | From Day 1 up to Day 121
The type of treatment-emergent Serious Adverse Events | From Day 1 up to Day 121

SECONDARY OUTCOMES:
AUC for each dose of REGN3048 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
AUC for each dose of REGN3051 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
AUC(0-infinity) for each dose of REGN3048 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
AUC(0-infinity) for each dose of REGN3051 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
CL for each dose of REGN3048 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
CL for each dose of REGN3051 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
CMAX for each dose of REGN3048 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
CMAX for each dose of REGN3051 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
K(e) for each dose of REGN3048 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
K(e) for each dose of REGN3051 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
t(1/2) for each dose of REGN3048 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
t(1/2) for each dose of REGN3051 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
The change from baseline of antibodies against REGN3048 and REGN3051 (anti-drug antibodies, ADA), as measured in serum using validated bridging assays | Day 121
The change from baseline of antibodies against REGN3048 and REGN3051 (anti-drug antibodies, ADA), as measured in serum using validated bridging assays | Day 57
TMAX for each dose of REGN3048 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
TMAX for each dose of REGN3051 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
V(ss) for each dose of REGN3048 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121
V(ss) for each dose of REGN3051 measured using validated Enzyme Linked Immunosorbent Assays (ELISAs) | From Day 1 up to Day 121

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global Cypress Clinical Pharmacology Unit, Cypress, California, United States